CLINICAL TRIAL: NCT00948896
Title: A Randomized Controlled Trial of Monthly Dihydroartemisinin-piperaquine Versus Monthly Sulfadoxine-pyrimethamine Versus Daily Trimethoprim-sulfamethoxazole Versus No Therapy for the Prevention of Malaria
Brief Title: Chemopreventive Therapy for Malaria in Ugandan Children
Acronym: PROMOTE-Chemop
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Grant Dorsey, M.D, Ph.D., Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H9926-33953; NIH P01HD059454; 2009-077 (Other: Makerere Univ Fac of Med Research and Ethics Committee); HS-580 (Other: Uganda National Council for Science and Tech); 686/ESR/NDA/DID-11/2009 (Other: Uganda National Drug Authority); H9926-33953 and 10-01489 (Other: UCSF Committee on Human Research)
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Malaria
Keywords: Chemoprevention; Uganda; Malaria; Trimethoprim-sulfamethoxazole; Sulfadoxine-pyrimethamine; Dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: trimethoprim-sulfamethoxazole (TS; TMP/SMX)
- 2 (Experimental)
  Interventions: Drug: sulfadoxine-pyrimethamine (SP)
- 3 (Experimental)
  Interventions: Drug: dihydroartemisinin-piperaquine (DP)
- 4 (No Intervention)

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole (TS; TMP/SMX) — daily dosing, 20mgTMP/100mgSMX tabs, 80mgTMP/400mgSMX tabs
  Arms: 1
Drug: sulfadoxine-pyrimethamine (SP) — monthly dosing given as a single dose, 500mg/25mg tabs
  Arms: 2
Drug: dihydroartemisinin-piperaquine (DP) — monthly dosing given once a day for 3 consecutive days, 40mg/320mg tabs
  Arms: 3

SUMMARY:
Young African children living in high transmission areas suffer the greatest burden of malaria. In most African countries, such as Uganda, the only current preventive measure against malaria in high transmission settings is the use of insecticide treated bednets (ITNs). Preliminary data show that even in the setting of ITN use, young children living in a high transmission setting suffer almost 4 episodes of clinical malaria per year, highlighting the need for new preventive strategies. Chemopreventive strategies offer a potential means of reducing the burden of malaria among young children living in a high transmission setting. This study will compare the efficacy and safety of 3 promising chemopreventive strategies (monthly dihydroartemisinin-piperaquine, monthly sulfadoxine-pyrimethamine, daily trimethoprim-sulfamethoxazole) with the current standard of no chemoprevention and will be conducted in two distinct patient populations: 1) HIV-unexposed children (HIV-uninfected children born to HIV-uninfected mothers) and 2) HIV-exposed children (HIV-uninfected children born to HIV-infected mothers). The intervention will begin in HIV-unexposed children when they reach 6 months of age, the time at which the incidence of malaria begins to increase, and will be continued until the children reach 24 months of age, which prior data suggest is when the incidence of malaria begins to decline due to the development of semi-immunity. In addition, study participants will be followed for one additional year following chemopreventive therapy to examine for "rebound" in the incidence of malaria following our intervention. HIV-exposed children will begin the intervention when they have completed breastfeeding and have been confirmed to remain HIV-uninfected. The intervention will continue until study participants reach 24 months of age and then the study participants will be followed for an additional year to examine for rebound in the incidence of malaria. It is anticipated that the results of this study will provide valuable comparative data on the effect of different chemopreventive strategies on malaria incidence in two distinct patient populations at high risk for malaria. In addition it is anticipated the results of this study will provide insight into the development of naturally acquired antimalarial immunity in the setting of chemopreventive therapy that will differ in terms of the drug regimens, the age at which the intervention is started, and the HIV status of the mothers.

DETAILED DESCRIPTION:
Convenience sampling will be used to enroll a cohort of 600 HIV-uninfected infants between the ages of 4-5 months of age according to the following strata based on the mother's HIV status: 1) 200 HIV-exposed infants born to HIV-infected mothers, and 2) 400 HIV-unexposed infants born to HIV-uninfected mothers. Potential study participants will be identified from the Tororo District Hospital Antenatal Clinic and surrounding clinics providing routine pediatric care. Potential study participants less than 6 months of age and their parents/guardians will be referred to our study clinic for screening. Eligible children will be enrolled when they reach 4-5 months of age and followed until the age of 36 months for all their routine medical care at our designated study clinic. All mother-child pairs will receive 2 long lasting ITNs at enrollment and, as available, a basic care package including a safe water vessel, multivitamins and condoms. HIV-unexposed children will be randomized to one of four chemoprevention arms when they reach 6 months of age. All HIV-exposed children born to HIV-infected mothers will be given TS prophylaxis and mothers will be encouraged to introduce food at 6 months of life and continue breastfeeding until 1 year of life, in accordance with Ugandan Ministry of Health (MOH) guidelines. HIV-exposed children will retested for HIV approximately every 60 days during breastfeeding and 6 weeks following cessation of breastfeeding. HIV-exposed children who remain HIV-uninfected following cessation of breastfeeding will be randomized to one of four chemoprevention arms. HIV-exposed children who test positive for HIV during the course of the study (those who seroconvert during breastfeeding) will be excluded from the study and referred for appropriate care.

During the follow-up period, all patients presenting to the clinic with a new episode of fever will undergo standard evaluation (history, physical examination and Giemsa-stained blood smear) for the diagnosis of malaria. Children diagnosed with uncomplicated malaria will be treated with AL and children diagnosed with complicated malaria will be treated with quinine in accordance with national guidelines. Response to antimalarial therapy will be assessed using standardized guidelines. All AL treatment failures occurring within 14 days of diagnosis will be treated with quinine in accordance with national guidelines. In the event that a patient fails quinine therapy, therapy will be repeated with quinine plus clindamycin. Patients with complicated malaria who have contraindications to giving quinine will be treated with parenteral artesunate. All episodes diagnosed more than 14 days after a previous episode will be considered new episodes for treatment purposes. After two years of age, patients with uncomplicated malaria will have follow up visits on the days Antimalarial drugs are administered only (Day 0, 1, and 2). Routine assessments will be performed in the study clinic approximately every 30 days. Routine assessments will include review of study protocol with parents/guardians of study participants, assessment for any outside medical care, assessment for adherence to assigned chemopreventive therapy, a focused history and physical examination and routine blood smears for the detection of asymptomatic parasitemia. Routine phlebotomy will be performed approximately every 120 days for all study participants for CBC, glucose and ALT measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 -5 months
2. Confirmed HIV status of biological mother
3. Negative HIV DNA PCR test at time of enrollment for infants born to HIV-infected mothers
4. Infants born to HIV-infected mothers must be breastfeeding
5. Residency within 30km of the study clinic
6. Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
7. Provision of informed consent by parent/guardian

Exclusion Criteria:

1. History of allergy or sensitivity to TS, SP, or DP
2. Active medical problem requiring in-patient evaluation at the time of screening
3. Intention of moving more that 30km from the study clinic during the follow-up period
4. Chronic medical condition (i.e. malignancy) requiring frequent medical attention
5. Living in the same household as a previously enrolled study participant
6. QTc interval > 450 msec
7. Other clinically significant ECG abnormalities such as arrhythmia, ischemia, or evidence of heart failure
8. Family history of Long QT syndrome
9. Current use of drugs that prolong the QT interval

Ages: 4 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2010-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V. Havlir, MD, Study Director — University of California, San Francisco; M. Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco; Moses R Kamya MBChB, MMed, MPH, Principal Investigator — Makerere University; IDRC
Locations (1):
- IDRC Research Clinic -Tororo District Hospital, Tororo, Uganda

REFERENCES:
- [Result] Osterbauer B, Kapisi J, Bigira V, Mwangwa F, Kinara S, Kamya MR, Dorsey G. Factors associated with malaria parasitaemia, malnutrition, and anaemia among HIV-exposed and unexposed Ugandan infants: a cross-sectional survey. Malar J. 2012 Dec 27;11:432. doi: 10.1186/1475-2875-11-432. PMID 23270614
- [Result] Ochong E, Tumwebaze PK, Byaruhanga O, Greenhouse B, Rosenthal PJ. Fitness Consequences of Plasmodium falciparum pfmdr1 Polymorphisms Inferred from Ex Vivo Culture of Ugandan Parasites. Antimicrob Agents Chemother. 2013 Sep;57(9):4245-4251. doi: 10.1128/AAC.00161-13. Epub 2013 Jun 24. PMID 23796921
- [Result] Marquez C, Okiring J, Chamie G, Ruel TD, Achan J, Kakuru A, Kamya MR, Charlebois ED, Havlir DV, Dorsey G. Increased morbidity in early childhood among HIV-exposed uninfected children in Uganda is associated with breastfeeding duration. J Trop Pediatr. 2014 Dec;60(6):434-41. doi: 10.1093/tropej/fmu045. Epub 2014 Aug 21. PMID 25145704
- [Result] Kamya MR, Kapisi J, Bigira V, Clark TD, Kinara S, Mwangwa F, Muhindo MK, Kakuru A, Aweeka FT, Huang L, Jagannathan P, Achan J, Havlir DV, Rosenthal PJ, Dorsey G. Efficacy and safety of three regimens for the prevention of malaria in young HIV-exposed Ugandan children: a randomized controlled trial. AIDS. 2014 Nov 28;28(18):2701-9. doi: 10.1097/QAD.0000000000000497. PMID 25493596
- [Result] Kapisi J, Bigira V, Clark T, Kinara S, Mwangwa F, Achan J, Kamya M, Soremekun S, Dorsey G. Efficacy and safety of artemether-lumefantrine for the treatment of uncomplicated malaria in the setting of three different chemopreventive regimens. Malar J. 2015 Feb 5;14:53. doi: 10.1186/s12936-015-0583-9. PMID 25652127
- [Result] Snyman K, Mwangwa F, Bigira V, Kapisi J, Clark TD, Osterbauer B, Greenhouse B, Sturrock H, Gosling R, Liu J, Dorsey G. Poor housing construction associated with increased malaria incidence in a cohort of young Ugandan children. Am J Trop Med Hyg. 2015 Jun;92(6):1207-13. doi: 10.4269/ajtmh.14-0828. Epub 2015 Apr 13. PMID 25870429
- [Result] Bigira V, Kapisi J, Clark TD, Kinara S, Mwangwa F, Muhindo MK, Osterbauer B, Aweeka FT, Huang L, Achan J, Havlir DV, Rosenthal PJ, Kamya MR, Dorsey G. Protective efficacy and safety of three antimalarial regimens for the prevention of malaria in young Ugandan children: a randomized controlled trial. PLoS Med. 2014 Aug 5;11(8):e1001689. doi: 10.1371/journal.pmed.1001689. eCollection 2014 Aug. PMID 25093754
- [Result] Sundell K, Jagannathan P, Huang L, Bigira V, Kapisi J, Kakuru MM, Savic R, Kamya MR, Dorsey G, Aweeka F. Variable piperaquine exposure significantly impacts protective efficacy of monthly dihydroartemisinin-piperaquine for the prevention of malaria in Ugandan children. Malar J. 2015 Sep 24;14:368. doi: 10.1186/s12936-015-0908-8. PMID 26403465
- [Result] Tumwebaze P, Conrad MD, Walakira A, LeClair N, Byaruhanga O, Nakazibwe C, Kozak B, Bloome J, Okiring J, Kakuru A, Bigira V, Kapisi J, Legac J, Gut J, Cooper RA, Kamya MR, Havlir DV, Dorsey G, Greenhouse B, Nsobya SL, Rosenthal PJ. Impact of antimalarial treatment and chemoprevention on the drug sensitivity of malaria parasites isolated from ugandan children. Antimicrob Agents Chemother. 2015;59(6):3018-30. doi: 10.1128/AAC.05141-14. Epub 2015 Mar 9. PMID 25753626
- See also: MU-UCSF Research Collaboration — http://www.muucsf.org/projects/chemo.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Convenience sampling was used to enroll a cohort of 600 infants 4-5 months of age from the Tororo District Hospital Maternal and Child Health clinic between June 2010 and July 2011.
Pre-assignment Details: Of the 400 HIV-unexposed infants, 7 were excluded prior to randomization for inability to comply with study protocol.
  Of the 200 HIV-exposed infants, 14 were excluded prior to randomization for the following reasons: 7 tested HIV positive; 3 unable to locate for > 60 days; 2 withdrew informed consent; 1 died; 1 unable to comply with protocol.
Groups:
- HIV-unexposed & No Chemoprevention: HIV-unexposed No chemoprevention was given
- HIV-unexposed & SP: HIV-unexposed sulfadoxine-pyrimethamine (SP): monthly dosing given as a single dose, 500mg/25mg tabs
- HIV-unexposed & TS: HIV-unexposed trimethoprim-sulfamethoxazole (TS; TMP/SMX): daily dosing, 20mgTMP/100mgSMX tabs, 80mgTMP/400mgSMX tabs
- HIV-unexposed & DP: HIV-unexposed dihydroartemisinin-piperaquine (DP): monthly dosing given once a day for 3 consecutive days, 40mg/320mg tabs
- HIV-exposed & no Chemoprevention: HIV-exposed No chemoprevention was given
- HIV-exposed & SP: HIV-exposed sulfadoxine-pyrimethamine (SP): monthly dosing given as a single dose, 500mg/25mg tabs
- HIV-exposed & TS: HIV-exposed trimethoprim-sulfamethoxazole (TS; TMP/SMX): daily dosing, 20mgTMP/100mgSMX tabs, 80mgTMP/400mgSMX tabs
- HIV-exposed & DP: HIV-exposed dihydroartemisinin-piperaquine (DP): monthly dosing given once a day for 3 consecutive days, 40mg/320mg tabs
Period: Randomization to 24 Months of Age
Arm/Group | HIV-unexposed & No Chemoprevention | HIV-unexposed & SP | HIV-unexposed & TS | HIV-unexposed & DP | HIV-exposed & no Chemoprevention | HIV-exposed & SP | HIV-exposed & TS | HIV-exposed & DP
Started | 98 | 98 | 99 | 98 | 46 | 46 | 47 | 47
Completed | 90 | 85 | 90 | 87 | 44 | 42 | 43 | 45
Not Completed | 8 | 13 | 9 | 11 | 2 | 4 | 4 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 4 | 4 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 2 | 5 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Moved out of Study Area | 0 | 3 | 3 | 1 | 0 | 2 | 0 | 0
Period: 24 Months of Age to 36 Months of Age
Arm/Group | HIV-unexposed & No Chemoprevention | HIV-unexposed & SP | HIV-unexposed & TS | HIV-unexposed & DP | HIV-exposed & no Chemoprevention | HIV-exposed & SP | HIV-exposed & TS | HIV-exposed & DP
Started | 90 | 85 | 90 | 87 | 44 | 42 | 43 | 45
Completed | 87 | 83 | 85 | 85 | 43 | 40 | 43 | 45
Not Completed | 3 | 2 | 5 | 2 | 1 | 2 | 0 | 0
Not completed — Death | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Moved out of Study Area | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Convenience sampling was used to enroll a cohort of 600 infants 4-5 mo of age from the Tororo District Hospital Maternal and Child Health Clinic between June 2010 and July 2011. The baseline characteristics were taken at enrollment.
Groups:
- HIV-unexposed & Monthly SP: HIV-unexposed sulfadoxine-pyrimethamine (SP): monthly dosing given as a single dose, 500mg/25mg tabs
- HIV-unexposed & Daily TS: HIV-unexposed trimethoprim-sulfamethoxazole (TS; TMP/SMX): daily dosing, 20mgTMP/100mgSMX tabs, 80mgTMP/400mgSMX tabs
- HIV-unexposed & Monthly DP: HIV-unexposed dihydroartemisinin-piperaquine (DP): monthly dosing given once a day for 3 consecutive days, 40mg/320mg tabs
- HIV-exposed & Monthly SP: HIV-exposed sulfadoxine-pyrimethamine (SP): monthly dosing given as a single dose, 500mg/25mg tabs
- HIV-exposed & Daily TS: HIV-exposed trimethoprim-sulfamethoxazole (TS; TMP/SMX): daily dosing, 20mgTMP/100mgSMX tabs, 80mgTMP/400mgSMX tabs
- HIV-exposed & Monthly DP: HIV-exposed dihydroartemisinin-piperaquine (DP): monthly dosing given once a day for 3 consecutive days, 40mg/320mg tabs
- Total: Total of all reporting groups
Arm/Group | HIV-unexposed & no Chemoprevention | HIV-unexposed & Monthly SP | HIV-unexposed & Daily TS | HIV-unexposed & Monthly DP | HIV-exposed & no Chemoprevention | HIV-exposed & Monthly SP | HIV-exposed & Daily TS | HIV-exposed & Monthly DP | Total
Number analyzed (Participants) | 98 | 98 | 99 | 98 | 46 | 46 | 47 | 47 | 579
Age, Continuous [Mean (Standard Deviation); unit: months] — Age in months at time of enrollment
  months | 5.4 (0.5) | 5.3 (0.5) | 5.4 (0.5) | 5.4 (0.5) | 4.8 (0.7) | 4.7 (0.7) | 4.8 (0.8) | 4.7 (0.8) | 5.2 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 48 | 52 | 22 | 21 | 27 | 25 | 287
  Male | 50 | 54 | 51 | 46 | 24 | 25 | 20 | 22 | 292
Slept under any bednet prior night [Number; unit: participants]
  Yes | 41 | 43 | 40 | 45 | 27 | 27 | 26 | 29 | 278
  No | 57 | 55 | 59 | 53 | 19 | 19 | 21 | 18 | 301
Slept under ITN prior night [Number; unit: participants]
  Yes | 27 | 30 | 27 | 29 | 22 | 24 | 19 | 22 | 200
  No | 71 | 68 | 72 | 69 | 24 | 22 | 28 | 25 | 379
Stunted [Number; unit: participants] — Length-for-age z-score <-2
  participants
    Yes | 10 | 11 | 6 | 4 | 6 | 7 | 6 | 7 | 57
    No | 88 | 87 | 93 | 94 | 40 | 39 | 41 | 40 | 522
Wasted [Number; unit: participants] — Weight-for-age Z-score < -2
  participants
    Yes | 4 | 7 | 7 | 5 | 0 | 4 | 1 | 4 | 32
    No | 94 | 91 | 92 | 93 | 46 | 42 | 46 | 43 | 547
Hemoglobin [Mean (Standard Deviation); unit: gm/dl] | 9.7 (1.4) | 9.6 (1.8) | 9.9 (1.5) | 9.5 (1.5) | 10.1 (1.2) | 10.0 (1.4) | 10.1 (1.1) | 10.5 (1.5) | 9.8 (1.5)
Positive thick blood smear [Number; unit: participants]
  Yes | 22 | 27 | 17 | 28 | 8 | 4 | 8 | 6 | 120
  No | 76 | 71 | 82 | 70 | 38 | 42 | 39 | 41 | 459
Taking TS prophylaxis [Number; unit: participants] — This measurement is only applicable for the HIV-exposed participants (n=186).
  participants
    Yes | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | 5 | 7 | 5 | 9 | NA — Total not calculated because data are not available (NA) in one or more arms.
    No | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | NA — Only applicable for HIV-exposed participants | 41 | 39 | 42 | 38 | NA — Total not calculated because data are not available (NA) in one or more arms.
Age at time of randomization [Median (Full Range); unit: months] | 6.0 [6.0 to 6.5] | 6.0 [6.0 to 6.5] | 6.0 [6.0 to 6.3] | 6.0 [6.0 to 6.5] | 10.0 [6.0 to 18.0] | 9.3 [6.5 to 18.8] | 11.6 [6.2 to 18.7] | 10.3 [6.5 to 20.0] | 6.0 [6.0 to 20.0]
Duration of follow-up [Median (Full Range); unit: days] | 547 [53 to 580] | 547 [63 to 550] | 547 [58 to 564] | 547 [7 to 569] | 427 [88 to 549] | 420 [127 to 524] | 346 [88 to 505] | 409 [31 to 535] | 546 [7 to 580]

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Any Adverse Events Defined as Severity Grade 3-4 That Are Possibly, Probably, or Definitely Related to Study Drugs
Description: NIH Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events published December, 2004
Time Frame: Time from randomization until 24 months of age
Measure: Number; unit: incidence per person-year at risk
Arm/Group | HIV-unexposed & no Chemoprevention | HIV-unexposed & Monthly SP | HIV-unexposed & Daily TS | HIV-unexposed & Monthly DP | HIV-exposed & no Chemoprevention | HIV-exposed & Monthly SP | HIV-exposed & Daily TS | HIV-exposed & Monthly DP
Number analyzed (Participants) | 98 | 98 | 99 | 98 | 46 | 46 | 47 | 47
incidence per person-year at risk
  All grade 3-4 adverse events | 1.159 | 1.415 | 0.914 | 0.611 | 1.214 | 1.478 | 0.659 | 0.678
  Grade 3-4 AEs possibly related to study drugs | NA — No study drugs taken. | 0.056 | 0.054 | 0.021 | NA — No study drugs taken. | 0 | 0.062 | 0.097
  All serious adverse events | 0.178 | 0.364 | 0.196 | 0.091 | 0.411 | 0.453 | 0.330 | 0.194
  Elevated Temperature | 0.542 | 0.546 | 0.393 | 0.323 | 0.431 | 0.532 | 0.206 | 0.174
  Anemia | 0.384 | 0.602 | 0.318 | 0.168 | 0.705 | 0.631 | 0.206 | 0.291
  Thrombocytopenia | 0.123 | 0.119 | 0.061 | 0.035 | 0 | 0.118 | 0 | 0.058
  Elevated aspartate aminotransferase | 0.048 | 0.056 | 0.041 | 0.021 | 0.039 | 0.020 | 0.041 | 0.039
  Elevated alanine aminotransferase | 0.027 | 0.028 | 0.027 | 0.021 | 0 | 0 | 0 | 0
  Neutropenia | 0.021 | 0.042 | 0.014 | 0.007 | 0 | 0 | 0 | 0
  Malnutrition | 0 | 0 | 0 | 0 | 0.020 | 0.020 | 0.021 | 0.039
Statistical Analysis 1: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly DP; Null Hypothesis: Within HIV-unexposed participants, there is no difference in the incidence of all grade 3-4 adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.0001, Negative Binomial Regression
Statistical Analysis 2: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly DP; Null Hypothesis: Within HIV-unexposed participants, there is no difference in the incidence of elevated temperature adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.01, Negative Binomial Regression — Monthly DP arm compared to No chemoprevention arm
Statistical Analysis 3: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly DP; Null Hypothesis: Within HIV-unexposed participants, there is no difference in the incidence of anemia adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.01, Negative Binomial Regression — Monthly DP arm compared to No chemoprevention arm
Statistical Analysis 4: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly DP; Null Hypothesis: Within HIV-unexposed participants, there is no difference in the incidence of thrombocytopenia adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.05, Negative Binomial Regression — Monthly DP arm compared to No chemoprevention arm
Statistical Analysis 5: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Monthly DP; Null Hypothesis: Within HIV-exposed participants, there is no difference in the incidence of all grade 3-4 adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.05, Negative Binomial Regression — Monthly DP arm compared with no chemoprevention arm
Statistical Analysis 6: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Monthly DP; Null Hypothesis: Within HIV-exposed participants, there is no difference in the incidence of anemia adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.05, Negative Binomial Regression — Monthly DP arm compared with no chemoprevention arm
Statistical Analysis 7: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Monthly DP; Null Hypothesis: Within HIV-exposed participants, there is no difference in the incidence of elevated temperature adverse events per PYAR between the control arm and the monthly DP arm; Test type: Superiority or Other; p < 0.05, Negative Binomial Regression — Monthly DP arm compared with the no chemoprevention arm
Statistical Analysis 8: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Daily TS; Null Hypothesis: Within HIV-exposed participants, there is no difference in the incidence of anemia adverse events per PYAR between the control arm and the daily TS arm; Test type: Superiority or Other; p < 0.01, Negative Binomial Regression — Daily TS arm compare with the no chemoprevention arm

2. Secondary Outcome: Rebound Incidence of Malaria Defined as the Number of Treatments for New Episodes of Malaria Per Time at Risk
Time Frame: 24 months to 36 months of age
Measure: Number; unit: Incidence per person year at risk
Arm/Group | HIV-unexposed & no Chemoprevention | HIV-unexposed & Monthly SP | HIV-unexposed & Daily TS | HIV-unexposed & Monthly DP | HIV-exposed & no Chemoprevention | HIV-exposed & Monthly SP | HIV-exposed & Daily TS | HIV-exposed & Monthly DP
Number analyzed (Participants) | 87 | 83 | 85 | 85 | 43 | 40 | 43 | 45
Incidence per person year at risk
  All incident episodes of malaria | 10.85 | 11.98 | 10.90 | 10.77 | 9.08 | 6.75 | 8.13 | 6.78
  Complicated malaria | 0.046 | 0.132 | 0.046 | 0 | 0.161 | 0.147 | 0.116 | 0.044
  All-cause hospital admissions | 0.046 | 0.452 | 0.091 | 0.023 | 0.459 | 0.318 | 0.186 | 0.089

3. Primary Outcome: Incident Malaria Cases Per Person Year at Risk in HIV-unexposed Participants
Description: The incidence of malaria, defined as the number of incident episodes per time at risk, during the period the intervention was given (6-24 mo of age). Treatments within 14d of a prior episode were not considered incident events. Time at risk was from the day following the initiation of study drugs to the last day of observation, minus 14 d after each treatment for malaria.
Time Frame: 6 to 24 months of age
Measure: Number; unit: Episode per person year at risk
Arm/Group | HIV-unexposed & no Chemoprevention | HIV-unexposed & Monthly SP | HIV-unexposed & Daily TS | HIV-unexposed & Monthly DP
Number analyzed (Participants) | 98 | 98 | 99 | 98
Episode per person year at risk
  6-24 mo. of Age | 6.95 | 6.73 | 5.21 | 3.02
  6-11 mo. of Age | 6.41 | 5.51 | 3.27 | 1.49
  12-24 mo. of Age | 7.24 | 7.41 | 6.32 | 3.88
Statistical Analysis 1: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly SP; The sample size was calculated to detect at least a 32% lower incidence of malaria in the DP arm compared to that in the TS arm. We assumed that the incidence of malaria would be 1.85 episodes per person-year with TS chemoprevention based on a prior cohort study in the same area, and thus we calculated that we would need to enroll 100 participants in each arm to detect our targeted protective efficacy with 80% power at 95% significance (two-sided), allowing for 10% loss to follow-up; Test type: Superiority or Other; p = 0.57, Negative Binomial Regression; Protective Efficacy (%) = 7, 95% CI 2-sided [-19 to 28] — The no chemoprevention arm is the reference group
Statistical Analysis 2: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Daily TS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.01, Negative Binomial Regression; Protective Efficacy (%) = 28, 95% CI 2-sided [7 to 44] — The no chemoprevention arm is the reference arm
Statistical Analysis 3: Comparison: HIV-unexposed & no Chemoprevention vs HIV-unexposed & Monthly DP; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Negative Binomial Regression; Protective Efficacy (%) = 58, 95% CI 2-sided [45 to 67] — The no chemoprevention arm is the reference arm

4. Primary Outcome: Incident Malaria Cases Per Person Year at Risk in HIV-exposed Participants
Description: The primary outcome was the incidence of malaria, defined as the number of incident episodes per time at risk, during the period the intervention was given. Treatments within 14 days of a prior episode were not considered incident events. Time at risk was from the day following the initiation of study drugs to the last day of observation, minus 14 days after each treatment for malaria.
Time Frame: Randomization to 24 months of age
Measure: Number; unit: Episodes per person year at risk
Arm/Group | HIV-exposed & no Chemoprevention | HIV-exposed & Monthly SP | HIV-exposed & Daily TS | HIV-exposed & Monthly DP
Number analyzed (Participants) | 46 | 46 | 47 | 47
Episodes per person year at risk
  Randomization - 24 mo. of Age | 6.28 | 4.50 | 2.86 | 1.83
  Randomization -16 mo. of Age | 5.42 | 3.72 | 1.70 | 0.90
  17-24 mo. of Age | 7.04 | 5.22 | 3.79 | 2.67
Statistical Analysis 1: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Monthly SP; We assumed that the incidence of malaria would be 1.85 episodes per person year with TS based on a prior cohort study in the same area, and thus, that we would need to enroll 50 participants in each arm to detect a reduction in the incidence of malaria in either the monthly SP or DP arms (two-sided significance level 0.05) compared with the daily TS arm of 48% or greater with 80% power at 95% significance (two-sided), allowing for 10% loss to follow-up; Test type: Superiority or Other; p = 0.065, Negative Binomial Regression; Protective Efficacy (%) = 9, 95% CI 2-sided [-35 to 38] — The no chemoprevention arm is the reference arm
Statistical Analysis 2: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Daily TS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, Negative Binomial Regression — Adjusted for age at randomization and incidence of malaria prior to randomization; Protective Efficacy (%) = 49, 95% CI 2-sided [23 to 66] — Adjusted for age at randomization and incidence of malaria prior to randomization. The no chemoprevention arm is the reference arm
Statistical Analysis 3: Comparison: HIV-exposed & no Chemoprevention vs HIV-exposed & Monthly DP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Negative Binomial Regression — Adjusted for age at randomization and incidence of malaria prior to randomization; Protective Efficacy (%) = 69, 95% CI 2-sided [53 to 80] — [estimate comment as in outcome 4, analysis 2]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected in the time period between randomization and when intervention was stopped (24 mo. of Age).
Arm/Group | HIV-unexposed & no Chemoprevention | HIV-unexposed & Monthly SP | HIV-unexposed & Daily TS | HIV-unexposed & Monthly DP | HIV-exposed & no Chemoprevention | HIV-exposed & Monthly SP | HIV-exposed & Daily TS | HIV-exposed & Monthly DP
Serious Adverse Events (participants affected / at risk) | 22/98 | 25/98 | 20/99 | 10/98 | 10/46 | 14/46 | 10/47 | 8/47
Other Adverse Events (participants affected / at risk) | 70/98 | 66/98 | 58/99 | 49/98 | 28/46 | 28/46 | 11/47 | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | HIV-unexposed & no Chemoprevention (N=98) | HIV-unexposed & Monthly SP (N=98) | HIV-unexposed & Daily TS (N=99) | HIV-unexposed & Monthly DP (N=98) | HIV-exposed & no Chemoprevention (N=46) | HIV-exposed & Monthly SP (N=46) | HIV-exposed & Daily TS (N=47) | HIV-exposed & Monthly DP (N=47)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 15 (19) | 20 (45) | 14 (20) | 4 (5) | 8 (19) | 11 (17) | 4 (6) | 5 (6)
Dehydration (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrolyte imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Elevated ALT (SGPT) (Hepatobiliary disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated AST (SGOT) (Hepatobiliary disorders) | 6 (7) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated temperature (Endocrine disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor feeding (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/46 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septicemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-unexposed & no Chemoprevention (N=98) | HIV-unexposed & Monthly SP (N=98) | HIV-unexposed & Daily TS (N=99) | HIV-unexposed & Monthly DP (N=98) | HIV-exposed & no Chemoprevention (N=46) | HIV-exposed & Monthly SP (N=46) | HIV-exposed & Daily TS (N=47) | HIV-exposed & Monthly DP (N=47)
Anemia (Blood and lymphatic system disorders) | 31 (39) | 28 (44) | 21 (28) | 17 (19) | 14 (18) | 11 (15) | 3 (4) | 7 (10)
Chills (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated ALT (SGPT) (Hepatobiliary disorders) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Elevated AST (SGOT) (Hepatobiliary disorders) | 5 (6) | 7 (8) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Elevated temperature (Endocrine disorders) | 53 (77) | 49 (75) | 41 (58) | 32 (46) | 17 (22) | 19 (27) | 9 (10) | 6 (8)
Hyperglycemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septicemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 7 (12) | 5 (8) | 5 (5) | 0 (0) | 5 (6) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes